CLINICAL TRIAL: NCT01333748
Title: Search Allelic Imbalance of Expression of BRCA Genes in Hereditary Risk of Breast and/or Ovarian Cancer
Acronym: EXSAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Dr Agnès HARDOUIN, Centre François BACLESSE
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EXSAL; 2009-A00833-54 (Registry Identifier: ID-RCB number)
Record Dates: First submitted 2011-04-04; First posted 2011-04-12 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
Keywords: breast cancer; ovarian cancer; BRCA 1 and BRCA 2
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Breast Neoplasms; Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients group (Experimental): Patients with ovarian and/or breast cancer
  Interventions: Genetic: blood collection
- control population (Other): control population without history of breast and/or ovarian cancer
  Interventions: Genetic: blood collection

INTERVENTIONS:
Genetic: blood collection — blood collection for research quantification of allelic expression in the gene BRCA1.
  Arms: patients group
Genetic: blood collection — blood collection for research quantification of allelic expression in the gene BRCA1.
  Arms: control population

SUMMARY:
The purpose of this study is to determine proportion of patients presented a search allelic imbalance of expression of genes BRCA 1 and 2 in population with hereditary breast and/or ovarian cancer risk and negative for deletion mutation BRCA 1 and 2 genes

ELIGIBILITY:
Inclusion Criteria:

For patients

* Women with breast cancer and / or ovarian cancer meet criteria suggestive of a hereditary predisposition
* Deleterious mutation of BRCA1 and BRCA2 sought and not highlighted
* Age ≥ 18 years
* Agreeing to participate in the study (a collection of signed informed consent)

For control population

* Women with no history of breast and / or ovarian cancer and no family history of breast and / or ovarian cancer among family members on the 1st and 2nd degree before age 50 for breast cancer and before 60 years for ovarian cancer
* Agreeing to participate in the study (a collection of signed informed consent)

Exclusion Criteria:

For patients:

* Patients with a known deleterious mutation in BRCA1 and BRCA2
* Patients do not meet criteria suggestive of a hereditary predisposition
* Persons deprived of liberty or under guardianship (including guardianship)

For control population:

* Males
* Personal or family history of breast and / or ovarian cancer (breast or ovarian cancer in their family experienced 1st and 2nd degree before age 50 for breast cancer before age 60 for cancer ovarian)
* Persons deprived of liberty or under guardianship (including guardianship)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
estimate the proportion of patients with allelic imbalance at the level of expression of BRCA1 | blood sample at baseline, no follow-up in this study
  The main objective of this study is to estimate the proportion of patients with allelic imbalance at the level of expression of BRCA1 in a population meeting the criteria suggestive of a hereditary predisposition to breast and / or ovarian cancer , and negative for deleterious mutations of BRCA 1 and BRCA 2.

SECONDARY OUTCOMES:
Study the variability of the measurement of the allelic expression depending on the position of SNPs | blood sample at baseline, no follow-up in this study
  Study the variability of the measurement of the allelic expression depending on the position of SNPs (Single Nucleotide Polymorphism) in the gene, in order to extend this research to variants of unknown significance whatever their position in the gene.
proportion of patients with allelic imbalance at the level of expression of the BRCA2 gene | blood sample at baseline, no follow-up in this study
  Estimate the proportion of patients with allelic imbalance at the level of expression of the BRCA2 gene in the same population.
Observe the possible effect of age | blood sample at baseline, no follow-up in this study
  The frequency of allelic imbalance of expression will be compared depending on the age of the witnesses in the control population. The potential effect of age on the presence or absence of allelic imbalance of expression will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès HARDOUIN, MD, Principal Investigator — Centre François Baclesse
Locations (6):
- France (6):
  - Dr Pascaline BERTHET, Caen, Caen
  - Centre Eugène MARQUIS, Rennes, Rennes
  - Centre Hospitalier, Cherbourg
  - CHU, Rennes
  - Centre Henri BECQUEREL, Rouen
  - CHU, Rouen